CLINICAL TRIAL: NCT02277769
Title: A Phase 3 Confirmatory Study Investigating the Efficacy and Safety of Dupilumab Monotherapy Administered to Adult Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: Study of Dupilumab (REGN668/SAR231893) Monotherapy Administered to Adult Patients With Moderate-to-Severe Atopic Dermatitis
Acronym: SOLO 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R668-AD-1416
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Two subcutaneous injections of Placebo (for Dupilumab) as a loading dose on Day 1 followed by a single injection once weekly (qw) from Week 1 to Week 15.
  Interventions: Drug: Placebo (for Dupilumab)
- Dupilumab 300 mg every 2 weeks (q2w) (Experimental): Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a placebo alternating with single 300 mg injection of Dupilumab qw from Week 1 to Week 15.
  Interventions: Drug: Dupilumab; Drug: Placebo (for Dupilumab)
- Dupilumab 300 mg qw (Experimental): Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a single 300 mg injection of Dupilumab qw from Week 1 to Week 15.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Subcutaneous injection alternated among the different quadrants of the abdomen, upper thighs and upper arms.
  Other Names: DUPIXENT®; REGN668; SAR231893
  Arms: Dupilumab 300 mg every 2 weeks (q2w); Dupilumab 300 mg qw
Drug: Placebo (for Dupilumab) — Subcutaneous injection alternated among the different quadrants of the abdomen, upper thighs and upper arms.
  Arms: Dupilumab 300 mg every 2 weeks (q2w); Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group study to confirm the efficacy and safety of Dupilumab monotherapy in adults with moderate-to-severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

1. Chronic AD that has been present for at least 3 years before the screening visit;
2. ≥10% body surface area (BSA) of AD involvement at the screening and baseline visits;
3. Documented recent history (within 6 months before the screening visit) of inadequate response to treatment with topical medications or for whom topical treatments are otherwise medically inadvisable (eg, because of important side effects or safety risks).

Exclusion Criteria:

1. Participation in a prior Dupilumab clinical study.
2. Treatment with an investigational drug within 8 weeks or within 5 half-lives (if known), whichever is longer, before the baseline visit;
3. Having used any of the following treatments within 4 weeks before the baseline visit, or any condition that, in the opinion of the investigator, is likely to require such treatment(s) during the first 4 weeks of study treatment:

   * Immunosuppressive/ immunomodulating drugs (eg, systemic corticosteroids, cyclosporine, mycophenolate-mofetil, IFN-γ, Janus kinase inhibitors, azathioprine, methotrexate, etc.)
   * Phototherapy for AD
4. Regular use (more than 2 visits per week) of a tanning booth/ parlor within 4 weeks of the screening visit;
5. Treatment with a live (attenuated) vaccine within 12 weeks before the baseline visit;
6. History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening;
7. Positive with hepatitis B surface antigen (HBsAg) or hepatitis C antibody at the screening visit;
8. Active chronic or acute infection requiring systemic treatment within 2 weeks before the baseline visit;
9. Known or suspected history of immunosuppression;
10. Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study;
11. Women unwilling to use adequate birth control, if of reproductive potential and sexually active.

Note: The information listed above is not intended to contain all considerations relevant to a participant's potential participation in this clinical trial therefore not all inclusion/ exclusion criteria are listed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 708 (Actual)
Dates: Start 2014-11-30 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2016-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (93):
- United States (53):
  - Anniston, Alabama
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Bakersfield, California
  - Costa Mesa, California
  - Fremont, California
  - Long Beach, California
  - Los Angeles, California
  - Orange, California
  - Roseville, California
  - Temecula, California
  - Trumbull, Connecticut
  - Miami, Florida
  - Oviedo, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Alpharetta, Georgia
  - Atlanta, Georgia
  - Columbus, Georgia
  - Buffalo Grove, Illinois
  - Plainfield, Indiana
  - West Des Moines, Iowa
  - Overland Park, Kansas
  - Rockville, Maryland
  - Washington Park, Maryland
  - Boston, Massachusetts
  - Farmington Hills, Michigan
  - Minneapolis, Minnesota
  - Plymouth, Minnesota
  - Saint Joseph, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Bozeman, Montana
  - Las Vegas, Nevada
  - Verona, New Jersey
  - Forest Hills, New York
  - New York, New York
  - Smithtown, New York
  - Chapel Hill, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Jenkintown, Pennsylvania
  - Greer, South Carolina
  - Arlington, Texas
  - Austin, Texas
  - Bellaire, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Richmond, Virginia
  - Seattle, Washington
- Canada (11):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Surrey, British Columbia
  - St. John's, Newfoundland and Labrador
  - Ajax, Ontario
  - Mississauga, Ontario
  - Oakville, Ontario
  - Ottawa, Ontario
  - Peterborough, Ontario
  - Richmond Hill, Ontario
  - Montreal, Quebec
- France (3):
  - Lille
  - Marseille
  - Nantes
- Germany (6):
  - Berlin
  - Bochum
  - Darmstadt
  - Friedrichshafen
  - Hamburg
  - Kiel
- Hong Kong, Hong Kong
- Italy (3):
  - Lucca
  - Pisa
  - Roma
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Poland (6):
  - Elblag
  - Gdansk
  - Katowice
  - Poznan
  - Torun
  - Warsaw
- South Korea (4):
  - Busan
  - Gyeonggi-do
  - Incheon
  - Seoul
- Stockholm, Sweden
- United Kingdom (2):
  - London
  - Plymouth

REFERENCES:
- [Result] Simpson EL, Bieber T, Guttman-Yassky E, Beck LA, Blauvelt A, Cork MJ, Silverberg JI, Deleuran M, Kataoka Y, Lacour JP, Kingo K, Worm M, Poulin Y, Wollenberg A, Soo Y, Graham NM, Pirozzi G, Akinlade B, Staudinger H, Mastey V, Eckert L, Gadkari A, Stahl N, Yancopoulos GD, Ardeleanu M; SOLO 1 and SOLO 2 Investigators. Two Phase 3 Trials of Dupilumab versus Placebo in Atopic Dermatitis. N Engl J Med. 2016 Dec 15;375(24):2335-2348. doi: 10.1056/NEJMoa1610020. Epub 2016 Sep 30. PMID 27690741
- [Derived] Langley RG, Gherardi G, Coleman A, Ardeleanu M, Rodriguez-Marco A, Levy S, Bansal A, Chen Z, Rossi AB, Shumel B, Khokhar FA. The Safety Data of Dupilumab for the Treatment of Moderate-to-Severe Atopic Dermatitis in Infants, Children, Adolescents, and Adults. Am J Clin Dermatol. 2025 Nov;26(6):981-1002. doi: 10.1007/s40257-025-00952-w. Epub 2025 Sep 24. PMID 40993471
- [Derived] Kamal MA, Kosloski MP, Lai CH, Partridge MA, Rajadhyaksha M, Kanamaluru V, Bansal A, Shabbir A, Shumel B, Ardeleanu M, Richards SM, Yan H, Xu CR, Rodriguez-Marco A, Xiao J, Khokhar FA, Gherardi G, Babilonia E, Maloney J, Mortensen E, Akinlade B, Braunstein N, Stahl N, Torri A, Davis JD, DiCioccio AT. Immunogenicity of dupilumab in adult and pediatric patients with atopic dermatitis. Front Immunol. 2024 Nov 11;15:1466372. doi: 10.3389/fimmu.2024.1466372. eCollection 2024. PMID 39588375
- [Derived] Silverberg JI, Lynde CW, Abuabara K, Patruno C, de Benedetto A, Zhang H, Thomas RB, Bego-Le-Bagousse G, Khokhar FA, Vakil J, Marco AR, Levit NA. Efficacy and Safety of Dupilumab Maintained in Adults >/= 60 Years of Age with Moderate-to-Severe Atopic Dermatitis: Analysis of Pooled Data from Four Randomized Clinical Trials. Am J Clin Dermatol. 2023 May;24(3):469-483. doi: 10.1007/s40257-022-00754-4. Epub 2023 Feb 20. PMID 36808602
- [Derived] Paller AS, Silverberg JI, Cork MJ, Guttman-Yassky E, Lockshin B, Irvine AD, Kim MB, Kabashima K, Chen Z, Lu Y, Bansal A, Rossi AB, Shabbir A. Efficacy and Safety of Dupilumab in Patients With Erythrodermic Atopic Dermatitis: A Post Hoc Analysis of 6 Randomized Clinical Trials. JAMA Dermatol. 2023 Mar 1;159(3):255-266. doi: 10.1001/jamadermatol.2022.6192. PMID 36723913
- [Derived] Silverberg JI, Boguniewicz M, Hanifin J, Papp KA, Zhang H, Rossi AB, Levit NA. Dupilumab Treatment in Adults with Moderate-to-Severe Atopic Dermatitis is Efficacious Regardless of Age of Disease Onset: a Post Hoc Analysis of Two Phase 3 Clinical Trials. Dermatol Ther (Heidelb). 2022 Dec;12(12):2731-2746. doi: 10.1007/s13555-022-00822-x. Epub 2022 Oct 21. PMID 36269503
- [Derived] Wechsler ME, Klion AD, Paggiaro P, Nair P, Staumont-Salle D, Radwan A, Johnson RR, Kapoor U, Khokhar FA, Daizadeh N, Chen Z, Laws E, Ortiz B, Jacob-Nara JA, Mannent LP, Rowe PJ, Deniz Y. Effect of Dupilumab on Blood Eosinophil Counts in Patients With Asthma, Chronic Rhinosinusitis With Nasal Polyps, Atopic Dermatitis, or Eosinophilic Esophagitis. J Allergy Clin Immunol Pract. 2022 Oct;10(10):2695-2709. doi: 10.1016/j.jaip.2022.05.019. Epub 2022 May 28. PMID 35636689
- [Derived] Armstrong A, Blauvelt A, Simpson EL, Smith CH, Herranz P, Kataoka Y, Seo SJ, Ferrucci SM, Chao J, Chen Z, Rossi AB, Shumel B, Tomondy P. Continued Treatment with Dupilumab is Associated with Improved Efficacy in Adults with Moderate-to-Severe Atopic Dermatitis Not Achieving Optimal Responses with Short-Term Treatment. Dermatol Ther (Heidelb). 2022 Jan;12(1):195-202. doi: 10.1007/s13555-021-00643-4. Epub 2021 Dec 13. PMID 34897582
- [Derived] Paller AS, Tan JKL, Bagel J, Rossi AB, Shumel B, Zhang H, Abramova A. IGAxBSA composite for assessing disease severity and response in patients with atopic dermatitis. Br J Dermatol. 2022 Mar;186(3):496-507. doi: 10.1111/bjd.20872. Epub 2022 Feb 25. PMID 34726270
- [Derived] Griffiths C, de Bruin-Weller M, Deleuran M, Fargnoli MC, Staumont-Salle D, Hong CH, Sanchez-Carazo J, Foley P, Seo SJ, Msihid J, Chen Z, Cyr SL, Rossi AB. Dupilumab in Adults with Moderate-to-Severe Atopic Dermatitis and Prior Use of Systemic Non-Steroidal Immunosuppressants: Analysis of Four Phase 3 Trials. Dermatol Ther (Heidelb). 2021 Aug;11(4):1357-1372. doi: 10.1007/s13555-021-00558-0. Epub 2021 Jun 18. PMID 34142350
- [Derived] Hamilton JD, Harel S, Swanson BN, Brian W, Chen Z, Rice MS, Amin N, Ardeleanu M, Radin A, Shumel B, Ruddy M, Patel N, Pirozzi G, Mannent L, Graham NMH. Dupilumab suppresses type 2 inflammatory biomarkers across multiple atopic, allergic diseases. Clin Exp Allergy. 2021 Jul;51(7):915-931. doi: 10.1111/cea.13954. Epub 2021 Jun 26. PMID 34037993
- [Derived] Boguniewicz M, Beck LA, Sher L, Guttman-Yassky E, Thaci D, Blauvelt A, Worm M, Corren J, Soong W, Lio P, Rossi AB, Lu Y, Chao J, Eckert L, Gadkari A, Hultsch T, Ruddy M, Mannent LP, Graham NMH, Pirozzi G, Chen Z, Ardeleanu M. Dupilumab Improves Asthma and Sinonasal Outcomes in Adults with Moderate to Severe Atopic Dermatitis. J Allergy Clin Immunol Pract. 2021 Mar;9(3):1212-1223.e6. doi: 10.1016/j.jaip.2020.12.059. Epub 2021 Jan 13. PMID 33453450
- [Derived] Silverberg JI, Simpson EL, Guttman-Yassky E, Cork MJ, de Bruin-Weller M, Yosipovitch G, Eckert L, Chen Z, Ardeleanu M, Shumel B, Hultsch T, Rossi AB, Hamilton JD, Orengo JM, Ruddy M, Graham NMH, Pirozzi G, Gadkari A. Dupilumab Significantly Modulates Pain and Discomfort in Patients With Atopic Dermatitis: A Post Hoc Analysis of 5 Randomized Clinical Trials. Dermatitis. 2021 Oct 1;32(1S):S81-S91. doi: 10.1097/DER.0000000000000698. PMID 33165005
- [Derived] Alexis AF, Rendon M, Silverberg JI, Pariser DM, Lockshin B, Griffiths CE, Weisman J, Wollenberg A, Chen Z, Davis JD, Li M, Eckert L, Gadkari A, Shumel B, Rossi AB, Graham NM, Ardeleanu M. Efficacy of Dupilumab in Different Racial Subgroups of Adults With Moderate-to-Severe Atopic Dermatitis in Three Randomized, Placebo-Controlled Phase 3 Trials. J Drugs Dermatol. 2019 Aug 1;18(8):804-813. PMID 31424712
- [Derived] Wollenberg A, Beck LA, Blauvelt A, Simpson EL, Chen Z, Chen Q, Shumel B, Khokhar FA, Hultsch T, Rizova E, Rossi AB, Graham NMH, Pirozzi G, Lu Y, Ardeleanu M. Laboratory safety of dupilumab in moderate-to-severe atopic dermatitis: results from three phase III trials (LIBERTY AD SOLO 1, LIBERTY AD SOLO 2, LIBERTY AD CHRONOS). Br J Dermatol. 2020 May;182(5):1120-1135. doi: 10.1111/bjd.18434. Epub 2019 Dec 1. PMID 31407311
- [Derived] Eichenfield LF, Bieber T, Beck LA, Simpson EL, Thaci D, de Bruin-Weller M, Deleuran M, Silverberg JI, Ferrandiz C, Folster-Holst R, Chen Z, Graham NMH, Pirozzi G, Akinlade B, Yancopoulos GD, Ardeleanu M. Infections in Dupilumab Clinical Trials in Atopic Dermatitis: A Comprehensive Pooled Analysis. Am J Clin Dermatol. 2019 Jun;20(3):443-456. doi: 10.1007/s40257-019-00445-7. PMID 31066001
- [Derived] Silverberg JI, Simpson EL, Ardeleanu M, Thaci D, Barbarot S, Bagel J, Chen Z, Eckert L, Chao J, Korotzer A, Rizova E, Rossi AB, Lu Y, Graham NMH, Hultsch T, Pirozzi G, Akinlade B. Dupilumab provides important clinical benefits to patients with atopic dermatitis who do not achieve clear or almost clear skin according to the Investigator's Global Assessment: a pooled analysis of data from two phase III trials. Br J Dermatol. 2019 Jul;181(1):80-87. doi: 10.1111/bjd.17791. Epub 2019 Apr 11. PMID 30791102
- [Derived] Simpson EL. Dupilumab Improves General Health-Related Quality-of-Life in Patients with Moderate-to-Severe Atopic Dermatitis: Pooled Results from Two Randomized, Controlled Phase 3 Clinical Trials. Dermatol Ther (Heidelb). 2017 Jun;7(2):243-248. doi: 10.1007/s13555-017-0181-6. Epub 2017 May 13. PMID 28503712

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 10 countries between 03 December 2014 and 21 January 2016. A total of 962 participants were screened in the study.
Pre-assignment Details: Out of 962 participants, 708 were randomized and 707 were treated in the study. Participants were randomized in 1:1:1 ratio to receive Dupilumab 300 mg once weekly (qw), Dupilumab 300 mg every 2 weeks (q2w) or Placebo qw.
Groups:
- Placebo: Two subcutaneous injections of Placebo (for Dupilumab) as a loading dose on Day 1 followed by a single injection qw from Week 1 to Week 15.
- Dupilumab 300 mg q2w: Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a placebo alternating with single 300 mg injection of Dupilumab qw from Week 1 to Week 15.
Period: Overall Study
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Started | 236 | 233 | 239
Treated | 235 | 233 | 239
Safety Population | 234 (1 participant received at least 1 injection of Dupilumab 300mg(analyzed in Dupilumab 300 mg q2w arm)) | 236 (3 participants (1 [placebo] + 2 [Dupilumab 300 mg qw arm]) analyzed in Dupilumab 300 mg q2w arm) | 237 (2 participants received fewer injections of Dupilumab 300 mg (analyzed in Dupilumab 300 mg q2w arm))
Completed | 190 | 220 | 221
Not Completed | 46 | 13 | 18
Not completed — Protocol Violation | 3 | 3 | 5
Not completed — Lack of Efficacy | 17 | 0 | 4
Not completed — Adverse Event | 14 | 2 | 4
Not completed — Other than specified above | 12 | 8 | 5

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw | Total
Number analyzed (Participants) | 236 | 233 | 239 | 708
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (14.09) | 36.9 (13.96) | 37.1 (14.51) | 37.1 (14.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 96 | 100 | 300
  Male | 132 | 137 | 139 | 408
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 12 | 27
  Not Hispanic or Latino | 219 | 218 | 220 | 657
  Unknown or Not Reported | 9 | 8 | 7 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 50 | 44 | 45 | 139
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 20 | 13 | 15 | 48
  White | 156 | 165 | 168 | 489
  More than one race | 3 | 5 | 7 | 15
  Unknown or Not Reported | 7 | 6 | 4 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  North and South America | 116 | 114 | 116 | 346
  Western Europe | 54 | 54 | 55 | 163
  Eastern Europe | 38 | 37 | 39 | 114
  Asia Pacific | 28 | 28 | 29 | 85
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: units on a scale] — The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
  units on a scale | 33.6 (14.31) | 31.8 (13.08) | 31.9 (12.70) | 32.4 (13.39)
Investigator's Global Assessment (IGA) Score [Mean (Standard Deviation); unit: units on a scale] — IGA was an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0= clear; 1= almost clear; 2= mild; 3= moderate; 4= severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear).
  units on a scale | 3.5 (0.50) | 3.5 (0.50) | 3.5 (0.50) | 3.5 (0.50)
Weekly Average of Peak Daily Pruritus Numerical Rating Scale (NRS) [Mean (Standard Deviation); unit: units on a scale] — Pruritus NRS scale is an assessment tool that is used to report the intensity of participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0= no itch; 10= worst itch imaginable]). Population: Number of participants analyzed = participants with available data for the baseline parameter.
  units on a scale
    number analyzed (Participants) | 235 | 232 | 238 | 705
    (all) | 7.5 (1.85) | 7.6 (1.60) | 7.5 (1.81) | 7.5 (1.76)
Body Surface Area (BSA) Involvement with AD [Mean (Standard Deviation); unit: percentage of body surface area] — Body surface area affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined.
  percentage of body surface area | 54.3 (23.06) | 52.7 (21.23) | 52.2 (21.51) | 53.1 (21.94)
SCORing Atopic Dermatitis (SCORAD) Score [Mean (Standard Deviation); unit: units on a scale] — SCORAD was a clinical tool for assessing the severity of AD developed by the European Task Force on Atopic Dermatitis (Severity scoring of atopic dermatitis: the SCORAD index). Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology (Basel) 186 (1): 23-31. 1993. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) were assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease). Population: Number of participants analyzed = participants with available data for the baseline parameter.
  units on a scale
    number analyzed (Participants) | 233 | 230 | 236 | 699
    (all) | 69.2 (14.91) | 67.2 (13.48) | 67.5 (13.10) | 68.0 (13.86)
Dermatology Life Quality Index (DLQI) Score [Mean (Standard Deviation); unit: units on a scale] — The DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life (QOL). The 10 questions assessed QOL over the past week, with an overall scoring of 0 (absent disease) to 30 (severe disease); a high score indicative of a poor QOL.
  units on a scale | 15.4 (7.69) | 15.4 (7.07) | 16.0 (7.33) | 15.6 (7.37)
Patient Oriented Eczema Measure (POEM) [Mean (Standard Deviation); unit: units on a scale] — The POEM was a 7-item questionnaire that assessed disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor quality of life [QOL]).
  units on a scale | 21.0 (5.94) | 20.8 (5.49) | 20.9 (5.59) | 20.9 (5.67)
Global Individual Signs Score (GISS) [Mean (Standard Deviation); unit: units on a scale] — Individual components of the AD lesions (erythema, infiltration/ papulation, excoriations, and lichenification) were rated globally (each assessed for the whole body, not by anatomical region) on a 4-point scale (0= none, 1= mild, 2= moderate and 3= severe) using the EASI severity grading criteria. Total score ranges from 0 (absent disease) to 12 (severe disease).
  units on a scale | 9.2 (1.78) | 9.0 (1.80) | 9.0 (1.75) | 9.1 (1.77)
Total Hospital Anxiety Depression Scale (HADS) [Mean (Standard Deviation); unit: units on a scale] — The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression. Cut-offs for identifying psychiatric distress has been reported as 7 to 8 for possible presence, 10 to 11 for probable presence, and 14 to 15 for severe anxiety or depression. Population: Number of participants analyzed = participants with available data for the baseline parameter.
  units on a scale
    number analyzed (Participants) | 231 | 227 | 233 | 691
    (all) | 13.7 (8.32) | 13.7 (7.52) | 14.6 (8.24) | 14.0 (8.04)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Score of "0" or "1" and Reduction From Baseline of ≥2 Points at Week 16
Description: IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear). Participants with IGA score of "0" or "1" and a reduction from baseline of ≥2 points at Week 16 were reported. Values after first rescue treatment were set to missing and participants with missing IGA scores at Week 16 were considered as non-responders.
Time Frame: Week 16
Population: Full analysis set included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 236 | 233 | 239
percentage of participants | 8.5 | 36.1 | 36.4
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 27.6, 95% CI 2-sided [20.46 to 34.69] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 27.9, 95% CI 2-sided [20.87 to 34.99] — Dupilumab 300 mg qw vs Placebo

2. Secondary Outcome: Percentage of Participants With Eczema Area and Severity Index-75 (EASI-75) (≥75% Improvement From Baseline) at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-75 responders were the participants who achieved ≥75% overall improvement in EASI score from baseline to Week 16. Values after first rescue treatment use were set to missing and participants with missing EASI score at Week 16 were considered as non-responders.
Time Frame: Week 16
Population: Full analysis set included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 236 | 233 | 239
percentage of participants | 11.9 | 44.2 | 48.1
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when the previous endpoint was statistically significant at 0.025 level. Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 32.3, 95% CI 2-sided [24.75 to 39.94] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 36.3, 95% CI 2-sided [28.69 to 43.81] — Dupilumab 300 mg qw vs Placebo

3. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥4 Points) of Weekly Average of Peak Daily Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 16
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Participants achieving a reduction of ≥4 points from baseline in weekly average of peak daily pruritus NRS score at Week 16 were reported. Values after first rescue treatment were set to missing and participants with missing peak NRS at Week 16 were considered as non-responders.
Time Frame: Baseline to Week 16
Population: Full analysis set (FAS) included all randomized participants. Here, number of participants analyzed = participants with baseline peak pruritus NRS ≥4.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 221 | 225 | 228
percentage of participants | 9.5 | 36.0 | 39.0
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 26.5, 95% CI 2-sided [19.13 to 33.87] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 29.5, 95% CI 2-sided [22.11 to 36.95] — Dupilumab 300 mg qw vs Placebo

4. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥3 Points) in Weekly Average of Peak Daily Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 16
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Participants achieving a reduction of ≥3 points from baseline in weekly average of peak daily pruritus NRS score at Week 16 were reported. Values after first rescue treatment were set to missing and participants with missing peak NRS at Week 16 were considered as non-responders.
Time Frame: Baseline to Week 16
Population: Full analysis set (FAS) included all randomized participants. Here, number of participants analyzed = participants with baseline peak pruritus NRS ≥3.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 226 | 231 | 234
percentage of participants | 12.8 | 50.6 | 49.1
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 37.8, 95% CI 2-sided [30.03 to 45.60] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 36.3, 95% CI 2-sided [28.56 to 44.06] — Dupilumab 300 mg qw vs Placebo

5. Secondary Outcome: Percent Change From Baseline in Weekly Average of Peak Pruritus Numerical Rating Scale (NRS) Score to Week 16
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]).
Time Frame: Baseline to Week 16
Population: Full analysis set (FAS) included all randomized participants. Here, number of participants analyzed = participants with available data for this endpoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 105 | 195 | 182
percent change | -18.1 (27.66) | -47.2 (28.50) | -50.9 (30.56)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -28.9, 95% CI 2-sided [-36.04 to -21.83] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; Least square (LS) mean difference = -32.8, 95% CI 2-sided [-40.20 to -25.49] — Dupilumab 300 mg qw vs Placebo

6. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥4 Points) of Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 4
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Participants achieving a reduction of ≥4 points from baseline in weekly average of peak daily pruritus NRS score at Week 4 were reported. Values after first rescue treatment were set to missing and participants with missing peak NRS at Week 4 were considered as non-responders.
Time Frame: Baseline to Week 4
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 221 | 225 | 228
percentage of participants | 6.3 | 22.7 | 27.6
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 16.3, 95% CI 2-sided [9.99 to 22.68] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 21.3, 95% CI 2-sided [14.66 to 27.93] — Dupilumab 300 mg qw vs Placebo

7. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥4 Points) of Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 2
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Participants achieving a reduction of ≥4 points from baseline in weekly average of peak daily pruritus NRS score at Week 2 were reported. Values after first rescue treatment were set to missing and participants with missing peak NRS at Week 2 were considered as non-responders.
Time Frame: Baseline to Week 2
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 221 | 225 | 228
percentage of participants | 0.9 | 10.7 | 12.7
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 9.8, 95% CI 2-sided [5.54 to 13.98] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 11.8, 95% CI 2-sided [7.31 to 16.32] — Dupilumab 300 mg qw vs Placebo

8. Secondary Outcome: Change From Baseline in Peak Daily Pruritus Numerical Rating Scale (NRS) Score to Week 16
Description: as for outcome 5
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 105 | 195 | 182
units on a scale | -1.41 (1.973) | -3.56 (2.258) | -3.87 (2.426)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -2.10, 95% CI 2-sided [-2.605 to -1.587] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -2.47, 95% CI 2-sided [-2.982 to -1.957] — Dupilumab 300 mg qw vs Placebo

9. Secondary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score to Week 16
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 105 | 197 | 181
percent change | -33.7 (33.45) | -69.6 (27.84) | -71.6 (27.08)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = -36.2, 95% CI 2-sided [-43.46 to -28.86] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -38.2, 95% CI 2-sided [-45.55 to -30.88] — Dupilumab 300 mg qw vs Placebo

10. Secondary Outcome: Percentage of Participants With Eczema Area and Severity Index-50 (EASI-50) (≥50% Improvement From Baseline) at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-50 responders were the participants who achieved ≥50% overall improvement in EASI score from baseline to Week 16. Values after first rescue treatment were set to missing and participants with missing EASI-50 scores at Week 16 were considered as non-responders.
Time Frame: Week 16
Population: Full analysis set (FAS) included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 236 | 233 | 239
percentage of participants | 22.0 | 65.2 | 61.1
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 43.2, 95% CI 2-sided [35.12 to 51.29] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 39.1, 95% CI 2-sided [30.92 to 47.19] — Dupilumab 300 mg qw vs Placebo

11. Secondary Outcome: Percentage of Participants With Eczema Area and Severity Index-90 (EASI-90) (≥90% Improvement From Baseline) at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-90 responders were the participants who achieved ≥90% overall improvement in EASI score from baseline to Week 16. Values after first rescue treatment were set to missing and participants with missing EASI-90 scores at Week 16 were considered as non-responders.
Time Frame: Week 16
Population: Full analysis set (FAS) included all randomized participants.
Measure: Number; unit: percentage of particpants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 236 | 233 | 239
percentage of particpants | 7.2 | 30 | 30.5
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 22.8, 95% CI 2-sided [16.09 to 29.59] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 23.3, 95% CI 2-sided [16.63 to 30.05] — Dupilumab 300 mg qw vs Placebo

12. Secondary Outcome: Change From Baseline in Percent Body Surface Area (BSA) to Week 16
Description: BSA affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined.
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of body surface area
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 105 | 197 | 181
percentage of body surface area | -14.48 (17.810) | -31.69 (19.614) | -32.97 (20.400)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -17.99, 95% CI 2-sided [-22.062 to -13.927] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -19.51, 95% CI 2-sided [-23.491 to -15.529] — Dupilumab 300 mg qw vs Placebo

13. Secondary Outcome: Percent Change From Baseline in the SCORing Atopic Dermatitis (SCORAD) Score to Week 16
Description: SCORAD is a clinical tool for assessing the severity of AD developed by the European Task Force on Atopic Dermatitis (Severity scoring of atopic dermatitis: the SCORAD index). Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology (Basel) 186 (1): 23-31. 1993. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 105 | 193 | 178
percent change | -22.7 (25.48) | -53.5 (25.23) | -56.0 (25.53)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -31.4, 95% CI 2-sided [-37.36 to -25.40] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -33.8, 95% CI 2-sided [-39.75 to -27.80] — Dupilumab 300 mg qw vs Placebo

14. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) to Week 16
Description: The DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life (QOL). The 10 questions assessed QOL over the past week, with an overall scoring of 0 (absent disease) to 30 (severe disease); a high score was indicative of a poor QOL.
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 105 | 197 | 181
units on a scale | -4.0 (5.75) | -9.7 (6.20) | -10.3 (6.75)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -5.7, 95% CI 2-sided [-6.86 to -4.47] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -5.9, 95% CI 2-sided [-7.10 to -4.72] — Dupilumab 300 mg qw vs Placebo

15. Secondary Outcome: Change From Baseline in Patient Oriented Eczema Measure (POEM) to Week 16
Description: The POEM is a 7-item questionnaire that assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor quality of life [QOL]).
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 104 | 196 | 181
units on a scale | -3.8 (6.07) | -10.7 (6.89) | -11.7 (7.13)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -7.0, 95% CI 2-sided [-8.36 to -5.57] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -8.0, 95% CI 2-sided [-9.36 to -6.64] — Dupilumab 300 mg qw vs Placebo

16. Secondary Outcome: Change From Baseline in Hospital Anxiety Depression Scale (HADS) to Week 16
Description: HADS is a fourteen item scale. Seven of the items relate to anxiety and seven items relate to depression. Each item on the questionnaire is scored from 0 (minimum score) - 3 (maximum score) and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression. Cut-offs for identifying psychiatric distress has been reported as 7 to 8 for possible presence, 10 to 11 for probable presence, and 14 to 15 for severe anxiety or depression.
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 103 | 191 | 175
units on a scale | -1.0 (4.44) | -5.2 (5.42) | -6.2 (6.01)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -4.2, 95% CI 2-sided [-5.34 to -3.09] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -4.9, 95% CI 2-sided [-6.04 to -3.81] — Dupilumab 300 mg qw vs Placebo

17. Secondary Outcome: Percent Change From Baseline in Global Individual Signs Score (GISS) to Week 16
Description: Individual components of the AD lesions (erythema, infiltration/ papulation, excoriations, and lichenification) were rated globally (each assessed for the whole body, not by anatomical region) on a 4-point scale (0= none, 1= mild, 2= moderate and 3= severe) using the EASI severity grading criteria. Total score ranges from 0 (absent disease) to 12 (severe disease).
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 105 | 197 | 181
percent change | -20.3 (25.03) | -47.5 (27.0) | -48.4 (27.29)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -27.7, 95% CI 2-sided [-33.73 to -21.70] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -28.9, 95% CI 2-sided [-35.03 to -22.74] — Dupilumab 300 mg qw vs Placebo

18. Secondary Outcome: Percent Change From Baseline in Weekly Average of Peak Daily Pruritus NRS Score to Week 2
Description: as for outcome 5
Time Frame: Baseline to Week 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 223 | 224 | 229
percent change | -6.3 (21.91) | -24.1 (21.22) | -21.2 (24.96)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -17.7, 95% CI 2-sided [-21.96 to -13.53] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -15.0, 95% CI 2-sided [-19.16 to -10.78] — Dupilumab 300 mg qw vs Placebo

19. Secondary Outcome: Percentage of Participants With Skin Infection Treatment Emergent Adverse Events (TEAEs) Requiring Systemic Treatment
Description: Treatment-emergent adverse events (TEAEs) were defined as AEs that developed or worsened or became serious during on-treatment period (time from the first dose of study drug up to the end of study [Week 28]). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs. Statistical significance in the hierarchical testing of secondary hypotheses was broken at this endpoint. Therefore, subsequent secondary efficacy endpoints were not tested for statistical significance.
Time Frame: Baseline up to Week 16
Population: Safety analysis set (SAF) which included all randomized participants who received any study drug, and was analyzed as treated.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 234 | 236 | 237
percentage of participants | 0 | 0 | 0

20. Secondary Outcome: Percentage of Participants With Treatment Emergent Serious Adverse Events (TESAEs) From Baseline Through Week 16
Description: Any untoward medical occurrence in a participant who received investigational medicinal product (IMP) was considered an AE without regard to possibility of causal relationship with this treatment. Treatment-emergent adverse events (TEAEs) were defined as AEs that developed or worsened or became serious during on-treatment period (time from the first dose of study drug up to the end of study [Week 28]). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs.
Time Frame: Baseline up to Week 16
Population: Safety analysis set which included all randomized participants who received any study drug, and was analyzed based on the treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 234 | 236 | 237
percentage of participants | 5.6 | 1.7 | 3.4

21. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) Leading to Treatment Discontinuation From Baseline Through Week 16
Description: as for outcome 20
Time Frame: Baseline up to Week 16
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 234 | 236 | 237
percentage of participants | 2.1 | 0.8 | 1.3

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Week 28) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent adverse events that developed/worsened during the 'on-treatment period' (time form the first dose of study drug up to the end of study [Week 28]). Analysis was performed on safety population.
Groups:
- Placebo: Participants exposed to Placebo (for Dupilumab) for 16 weeks (mean exposure of 14 weeks)
- Dupilumab 300 mg q2w: Participants exposed to Dupilumab 300 mg alternating with placebo qw for 16 weeks (mean exposure of 15 weeks).
- Dupilumab 300 mg qw: Participants exposed to Dupilumab 300 mg qw for 16 weeks (mean exposure of 15 weeks).
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
All-Cause Mortality (participants affected / at risk) | 0/234 | 3/236 | 1/237
Serious Adverse Events (participants affected / at risk) | 16/234 | 6/236 | 9/237
Other Adverse Events (participants affected / at risk) | 109/234 | 84/236 | 90/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=234) | Dupilumab 300 mg q2w (N=236) | Dupilumab 300 mg qw (N=237)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Septic embolus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Tetany (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxic-Ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Schizophrenia, paranoid type (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 6 (8) | 0 (0) | 1 (1)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=234) | Dupilumab 300 mg q2w (N=236) | Dupilumab 300 mg qw (N=237)
Injection site reaction (General disorders) | 15 (17) | 32 (58) | 31 (84)
Nasopharyngitis (Infections and infestations) | 25 (26) | 23 (25) | 22 (26)
Headache (Nervous system disorders) | 12 (20) | 18 (29) | 23 (50)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 82 (136) | 34 (39) | 39 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not less than 45 days prior to submission for publication or presentation, the Institution shall, or cause the Principal Investigator to, provide the Sponsor with a copy of the Manuscript. The Institution shall consider in good faith any comments from the Sponsor regarding the content, and shall delete Confidential Information upon written request of the Sponsor. At the Sponsor's request, the Institution shall delay publication for an additional 60 days to allow patent applications to be filed.